CLINICAL TRIAL: NCT05071859
Title: Genetic Overlap Between Anomalies and Cancer in Kids in the Children's Oncology Group: The COG GOBACK Study
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AEPI19N1
Record Dates: First submitted 2021-09-28; First posted 2021-10-08 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Congenital Anomaly; Pediatric Cancer
Keywords: Congenital Anomaly
MeSH Terms: conditions — Congenital Abnormalities; Neoplasms | interventions — Whole Genome Sequencing

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva, germline, tumor samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GOBACK: The patient must have been diagnosed with cancer at ≤25 years of age and have been diagnosed with one or more congenital anomalies reported through the APEC14B1 registry intake data. For all patients in APEC14B1 with self-reported congenital anomalies the investigators will: 1) recruit cases; 2) administer the GOBACK Study questionnaire; 3) collect biological samples for sequencing; and 4) obtain medical records to verify anomalies. Medical records will be used to validate self-reported congenital anomalies and is a crucial step prior to sequencing. Additionally, the investigators will be able to identify those with well-established cancer predisposition syndromes that involve congenital anomalies, such as WAGR syndrome.
  Interventions: Other: Whole Genome Sequencing; Other: Questionnaire Administration; Other: Biospecimen collection; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Whole Genome Sequencing — Saliva collection and request for banked blood and tumor samples for sequencing
Other: Questionnaire Administration — Study questionnaire will include modules that collect information on maternal reproductive history, exposure to known teratogens, medical history, and previous genetic testing.
Other: Biospecimen collection — Saliva collection and request for banked blood and tumor samples for sequencing and biomarker analysis
Other: Laboratory Biomarker Analysis — Saliva collection and request for banked blood and tumor samples for biomarker analysis

SUMMARY:
One of the strongest risk factors for cancer in children and adolescents is being born with a congenital anomaly. In fact, data from registry linkage studies imply that 10-15% of childhood cancer risk could be attributable to having a congenital anomaly. As an estimated 10 million children worldwide are born with a congenital anomaly per year, the public health implications of identifying why some of these children develop cancer are thus substantial. While these studies have been informative, registry data alone offers no possibility of molecular or sequencing studies to identify the specific genetic basis underlying the co-occurrence of anomalies and cancer susceptibility. Therefore, the investigators developed the first phase of the Genetic Overlap Between Anomalies and Cancer in Kids (GOBACK) Study to address these limitations. Using data from birth defects and cancer registries from four states, the investigators identified numerous novel specific anomaly-cancer associations. In the GOBACK Study the investigators identified an increase in cancer risk among children with any chromosomal abnormality and any non-chromosomal birth defect. Additionally, children with congenital anomalies developed a variety of cancers, therefore the investigators propose to evaluate a range of cancers among children with congenital anomalies. By pooling registry data across four states in the GOBACK Study, the investigators found that children with non-chromosomal birth defects have a significantly elevated risk of several childhood cancers. Notably several of these congenital anomalies are not characteristic of known cancer predisposition syndromes. Therefore, our preliminary studies lay the framework for this application. The objectives of the current study are to (1) interrogate the genomes of children with co-occurring non-chromosomal congenital anomalies and cancer enrolled in Project:EveryChild to identify genetic features associated with these combined phenotypes, and (2) verify congenital anomalies and determine the phenotypic spectrum among children with cancer enrolled in Project:EveryChild with self-reported congenital anomalies ("deep phenotyping"). For this study the investigators will utilize Project:EveryChild to identify, contact, and enroll case-parent trios for children with co-occurring non-chromosomal congenital anomalies and cancers. From each enrolled family the investigators e will collect DNA from the affected case and one or both biological parents to comprise each case-parent trio. The investigators will include siblings if available. The investigators will also characterize case-parent trios based on demographic and clinical characteristics utilizing information collected via self-administered questionnaires and medical records. Ultimately the findings from this study could lead to 1) determining the potential genetic mechanisms that underlie these co-occurring conditions; 2) improving cancer risk-management strategies among children with birth defects; and 3) identifying the role congenital anomalies play in outcomes and survivorship among children diagnosed with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

1.1 Primary Aim Interrogate the genomes of children with co-occurring non-chromosomal congenital anomalies and cancer enrolled in Project:EveryChild to identify genetic features associated with these combined phenotypes.

1.2 Secondary Aim Verify congenital anomalies and determine the phenotypic spectrum among children with cancer enrolled in Project:EveryChild with self-reported congenital anomalies ("deep phenotyping").

ELIGIBILITY:
Inclusion Criteria:

* The patient must have been diagnosed with cancer at ≤25 years of age and have been diagnosed with one or more congenital anomalies reported through the APEC14B1 registry intake data. All types of non-syndromic birth defects and all types of cancers are eligible, regardless of patient vital status.

The patient must be enrolled on APEC14B1 with consent to future contact and registered with COG by a North American member institution. Note: (history of) treatment on a COG therapeutic trial is not required.

Language: English, French, or Spanish speaking.

The patient may participate regardless of the availability of biological parent(s).

Exclusion Criteria:

* Patients with a self-reported genetic syndrome as identified in the APEC14B1 Registry are not eligible.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patient must have been diagnosed with cancer at ≤25 years of age and have been diagnosed with one or more congenital anomalies reported through the APEC14B1 registry intake data. All types of non-syndromic birth defects and all types of cancers are eligible, regardless of patient vital status.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Interrogate the genomes of children with co-occurring non-chromosomal congenital anomalies and cancer enrolled in Project:EveryChild to identify genetic features associated with these combined phenotypes. | Up to 5 years
  Analyze de novo single-nucleotide variants (SNVs), copy number variants (CNVs), and insertions/deletions (INDELs) obtained through whole-genome sequencing of co-occurring non-chromosomal congenital anomalies and cancer case-parent trios, which are necessary to identify genes with de novo mutations. The investigators plan to enroll a maximum of 1,000 case-parent trios. For individuals on COG therapeutic studies, no treatment outcomes would be requested or reported as part of this study.

SECONDARY OUTCOMES:
Verify congenital anomalies and determine the phenotypic spectrum among children with cancer enrolled in Project:EveryChild with self-reported congenital anomalies (deep phenotyping). | Up to 5 years
  The primary analyses of data generated in this secondary aim will be descriptive in nature. The objective will largely be to verify congenital anomalies and determine the phenotypic spectrum of children with congenital anomalies and cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine/ Dan L Duncan Comprehensive Cancer Center, Houston, Texas, United States